CLINICAL TRIAL: NCT07364006
Title: Evaluation of Accuracy in Fully Guided Dental Implant Surgery Using 3D-Printed Surgical Guides Without Metal Sleeves: A Split-Mouth In Vivo Study
Brief Title: Accuracy of Metal Sleeve-Free Fully Guided Implant Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Miguel Gómez Polo, Associate Professor of conservative dentistry and prosthodontics, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 24/764-E
Record Dates: First submitted 2026-01-10; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Edentulism
Keywords: Guided implant surgery; Dental implants; Surgical guide accuracy; Metal sleeve-free surgical guides; 3D-printed surgical guides

STUDY DESIGN:
Intervention Model Description: Split-mouth design with intraindividual comparison of two drilling channel diameters using metal sleeve-free surgical guides.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Drilling Diameter (Experimental): Implant placement using metal sleeve-free 3D-printed surgical guides with a standard drilling channel diameter (4.85 mm).
  Interventions: Device: Standard Drilling Channel Metal Sleeve-Free Surgical Guide
- Reduced Drilling Diameter (Experimental): Implant placement using metal sleeve-free 3D-printed surgical guides with a reduced drilling channel diameter (4.83 mm).
  Interventions: Device: Reduced drilling channel Metal Sleeve-Free Surgical Guide

INTERVENTIONS:
Device: Standard Drilling Channel Metal Sleeve-Free Surgical Guide — Fully guided dental implant surgery performed using 3D-printed surgical guides without metal sleeves. The guides are designed based on virtual implant planning and used to place dental implants with a standard drilling channel diameter in a split-mouth design.
  Arms: Standard Drilling Diameter
Device: Reduced drilling channel Metal Sleeve-Free Surgical Guide — Fully guided dental implant surgery performed using 3D-printed surgical guides without metal sleeves. The guides are designed based on virtual implant planning and used to place dental implants with reduced drilling channel diameter in a split-mouth design.
  Arms: Reduced Drilling Diameter

SUMMARY:
This clinical trial aims to evaluate the in vivo accuracy of fully guided dental implant surgery using 3D-printed surgical guides without metal sleeves. The study is designed as a split-mouth clinical trial and will be conducted in partially or fully edentulous adult patients requiring complete-arch rehabilitation with dental implants.

The primary objective of the study is to assess the accuracy of implant placement by comparing the virtually planned implant positions with the actual clinical positions achieved after guided surgery. Accuracy will be evaluated by analyzing linear and angular deviations between planned and placed implants.

Participants will undergo a fully guided implant placement procedure using metal sleeve-free surgical guides. Two different drilling channel diameters (standard and reduced) will be randomly assigned in a split-mouth manner. Postoperative intraoral scans and cone-beam computed tomography (CBCT) scans with scan bodies will be obtained to register the final implant positions.

The planned and achieved implant positions will be compared using three-dimensional analysis software to quantify deviations and determine whether the use of metal sleeve-free guides and reduced drilling diameters influences implant placement accuracy.

DETAILED DESCRIPTION:
Background. Computer-guided implant surgery is associated with a known loss of accuracy when compared with virtual implant planning, due to the influence of multiple clinical and technical factors. Deviations between planned and actual implant positions remain a relevant issue in guided implant surgery. Accuracy is commonly assessed by comparing virtually planned implant positions with postoperative implant positions using linear and angular deviation measurements. From a clinical perspective, improving the accuracy of guided implant placement is particularly relevant in complete-arch rehabilitations, where small deviations may affect prosthetic fit and clinical outcomes. Metal sleeves incorporated into surgical guides may contribute to mechanical tolerance between the drilling instrument and the guide, and reducing this tolerance could potentially improve accuracy.

Justification. Despite the widespread use of guided implant surgery, limited in vivo evidence exists regarding the effect of eliminating metal sleeves from surgical guides on implant placement accuracy. Additionally, the influence of reducing the drilling channel diameter on implant deviation relative to virtual planning has not been sufficiently evaluated. This study aims to determine whether the elimination of metal sleeves and the reduction of drilling channel diameter improve the accuracy of guided implant surgery. The findings may help clarify whether the use of metal sleeves is necessary and whether reducing the drilling channel diameter compared with manufacturer standards may decrease implant deviation by minimizing the gap between the drill and the guide.

Study Design. This study is designed as a prospective, single-center, interventional split-mouth clinical trial. An intraindividual comparison will be performed between two guided surgery conditions within the same patient.

Participants. The study population will consist of 15 partially or fully edentulous patients requiring fixed complete-arch rehabilitation with dental implants. Eligible participants will be patients classified as ASA I or II. Patients classified as ASA III or IV will be excluded. All participants will be required to meet the predefined inclusion criteria, none of the exclusion criteria, and will be required to provide written informed consent prior to participation.

Intervention. Virtual implant planning will be performed using guided surgery software by aligning DICOM data from cone-beam computed tomography scans with STL files of the maxillae obtained through intraoral scanning. A virtual diagnostic wax-up of the immediate-loading provisional restoration will be created to guide prosthetically driven implant planning. Following virtual planning, two drilling conditions will be randomly assigned in a split-mouth manner. On one side, drilling channels will be designed with the standard diameter recommended by the manufacturer for use with metal sleeves (4.85 mm). On the contralateral side, drilling channels will be designed with a reduced diameter of 4.83 mm. Surgical guides will be digitally designed, exported as STL files, and fabricated using three-dimensional printing technology with biocompatible surgical guide resin at a resolution of 35 microns. The guides will be sterilized in an autoclave at 134 °C for 5 minutes. Dental implants will be placed using the guided surgical templates.

Outcomes Assessment. After implant placement, postoperative intraoral scans with scan bodies will be obtained, and cone-beam computed tomography scans with scan bodies will be performed following a standardized imaging protocol. The planned and postoperative datasets will be compared to evaluate differences between virtual implant planning and actual implant placement. Measurements will be performed using reverse engineering software to calculate linear and angular deviations between planned and placed implants.

Statistical Analysis. Once data collection is completed, statistical analysis will be performed. Data normality will be assessed, and a chi-square test will be used to evaluate differences between the study conditions.

ELIGIBILITY:
Inclusion Criteria:

* Partially or fully edentulous patients requiring fixed complete-arch rehabilitation with dental implants.
* Patients classified as ASA I or ASA II.
* Adult patients aged 18 years or older.
* Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Patients classified as ASA III or ASA IV.
* Patients with medical conditions that contraindicate dental implant surgery.
* Inability or unwillingness to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Drilling Channel Diameter on Implant Placement Accuracy | Immediately after implant placement
  Implant placement accuracy will be compared between implants placed using fully guided surgical guides with a standard drilling channel diameter (4.85 mm) and those placed using a reduced drilling channel diameter (4.83 mm). Linear deviations at the coronal and apical implant levels, as well as angular deviations of the implant axis, relative to the virtual implant planning will be measured to determine whether differences in accuracy exist between both drilling conditions.

SECONDARY OUTCOMES:
Deviation Between Planned and Actual Implant Positions | Immediately after implant placement
  The linear and angular deviations between the virtually planned implant positions and the actual implant positions achieved after fully guided implant surgery will be evaluated to describe overall implant placement accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ballesteros, DDs, MSc, Principal Investigator — Universidad Complutense de Madrid Juan Ballesteros- Martinez, DDs, MSc; Miguel A Gómez Polo, DDS, PhD, Study Chair — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gomez-Polo M, Ballesteros J, Padilla PP, Pulido PP, Revilla-Leon M, Ortega R. Merging intraoral scans and CBCT: a novel technique for improving the accuracy of 3D digital models for implant-supported complete-arch fixed dental prostheses. Int J Comput Dent. 2021 Jun 4;24(2):117-123. PMID 34085497
- [Background] Chen Z, Li J, Ceolin Meneghetti P, Galli M, Mendonca G, Wang HL. Does guided level (fully or partially) influence implant placement accuracy at post-extraction sockets and healed sites? An in vitro study. Clin Oral Investig. 2022 Aug;26(8):5449-5458. doi: 10.1007/s00784-022-04512-y. Epub 2022 May 2. PMID 35499656
- [Background] Pessoa R, Siqueira R, Li J, Saleh I, Meneghetti P, Bezerra F, Wang HL, Mendonca G. The Impact of Surgical Guide Fixation and Implant Location on Accuracy of Static Computer-Assisted Implant Surgery. J Prosthodont. 2022 Feb;31(2):155-164. doi: 10.1111/jopr.13371. Epub 2021 May 10. PMID 33904640
- [Background] Shah NP, Khanna A, Pai AR, Sheth VH, Raut SR. An evaluation of virtually planned and 3D-printed stereolithographic surgical guides from CBCT and digital scans: An in vitro study. J Prosthet Dent. 2022 Sep;128(3):436-442. doi: 10.1016/j.prosdent.2020.12.035. Epub 2021 Feb 12. PMID 33583616
- [Background] El Kholy K, Janner SFM, Schimmel M, Buser D. The influence of guided sleeve height, drilling distance, and drilling key length on the accuracy of static Computer-Assisted Implant Surgery. Clin Implant Dent Relat Res. 2019 Feb;21(1):101-107. doi: 10.1111/cid.12705. Epub 2018 Dec 27. PMID 30589502
- [Background] Hernandez-Margarit P, Palacios-Banuelos R, Roig M, Altuna P, Blasi A. Digital workflow for designing an interim implant-supported restoration with an optimal emergence profile in an open-source software program. J Prosthet Dent. 2024 Nov;132(5):857-862. doi: 10.1016/j.prosdent.2022.10.013. Epub 2022 Dec 6. PMID 36494239
- [Background] Derksen W, Wismeijer D, Flugge T, Hassan B, Tahmaseb A. The accuracy of computer-guided implant surgery with tooth-supported, digitally designed drill guides based on CBCT and intraoral scanning. A prospective cohort study. Clin Oral Implants Res. 2019 Oct;30(10):1005-1015. doi: 10.1111/clr.13514. Epub 2019 Sep 9. PMID 31330566
- [Background] Adams CR, Ammoun R, Deeb GR, Bencharit S. Influence of Metal Guide Sleeves on the Accuracy and Precision of Dental Implant Placement Using Guided Implant Surgery: An In Vitro Study. J Prosthodont. 2023 Jan;32(1):62-70. doi: 10.1111/jopr.13503. Epub 2022 Mar 22. PMID 35257456
- [Background] Abduo J, Lau D. Effect of Manufacturing Technique on the Accuracy of Surgical Guides for Static Computer-Aided Implant Surgery. Int J Oral Maxillofac Implants. 2020 Sep/Oct;35(5):931-938. doi: 10.11607/jomi.8186. PMID 32991643
- [Background] Henprasert P, Dawson DV, El-Kerdani T, Song X, Couso-Queiruga E, Holloway JA. Comparison of the Accuracy of Implant Position Using Surgical Guides Fabricated by Additive and Subtractive Techniques. J Prosthodont. 2020 Jul;29(6):534-541. doi: 10.1111/jopr.13161. Epub 2020 May 6. PMID 32147893
- [Background] Putra RH, Yoda N, Astuti ER, Sasaki K. The accuracy of implant placement with computer-guided surgery in partially edentulous patients and possible influencing factors: A systematic review and meta-analysis. J Prosthodont Res. 2022 Jan 11;66(1):29-39. doi: 10.2186/jpr.JPR_D_20_00184. Epub 2021 Jan 26. PMID 33504723
- [Background] Oh KC, Park JM, Shim JS, Kim JH, Kim JE, Kim JH. Assessment of metal sleeve-free 3D-printed implant surgical guides. Dent Mater. 2019 Mar;35(3):468-476. doi: 10.1016/j.dental.2019.01.001. Epub 2019 Jan 23. PMID 30685109
- [Background] Kernen F, Kramer J, Wanner L, Wismeijer D, Nelson K, Flugge T. A review of virtual planning software for guided implant surgery - data import and visualization, drill guide design and manufacturing. BMC Oral Health. 2020 Sep 10;20(1):251. doi: 10.1186/s12903-020-01208-1. PMID 32912273